CLINICAL TRIAL: NCT02678572
Title: A Single-arm, Multi-Center, Open-Label Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Melphalan/HDS Treatment in Patients With Hepatic-Dominant Ocular Melanoma
Brief Title: Percutaneous Hepatic Perfusion in Patients With Hepatic-dominant Ocular Melanoma
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Delcath Systems Inc. (Industry)
Collaborators: IQVIA Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHP-OCM-301A
Record Dates: First submitted 2016-02-01; First posted 2016-02-10 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Melanoma, Ocular
Keywords: uveal liver PHP hepatic perfusion chemosaturation Delcath
MeSH Terms: conditions — Uveal Melanoma | interventions — Melphalan

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single-arm, open-label study to evaluate the efficacy and safety of Melphalan/HDS in patients with hepatic dominant metastatic ocular melanoma. The study will be conducted at approximately 40 centers in the United States and Europe.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melphalan/HDS (Experimental): 3 mg/kg ideal body weight of melphalan for infusion administered directly to the liver via percutaneous hepatic perfusion (PHP) over 30 minutes followed by a 30 minute washout. Treatment cycles are to be repeated every 6-8 weeks until disease progression.
  Interventions: Combination Product: Melphalan/HDS

INTERVENTIONS:
Combination Product: Melphalan/HDS — Melphalan (3 mg/kg IBW) with Hepatic Device System (HDS)
  Other Names: Alkeran

SUMMARY:
This study will evaluate patients who have melanoma that has spread from the eye to the liver: Patients in the study will be treated with Melphalan/HDS up to 6 total treatment, and will be followed until death. This study will evaluate the safety and effects of the treatment on how long patients live and how long it takes for the cancer to advance or respond to the treatment.

DETAILED DESCRIPTION:
The study will consist of 3 phases: a screening phase, treatment phase, and follow-up phase.

Screening Phase: Screening assessments will be conducted within 28 days prior to the eligibility date to determine each patient's overall eligibility and baseline characteristics. These assessments will include medical history, physical examination, Eastern Cooperative Oncology Group (ECOG) performance status (PS), 12 lead electrocardiogram (ECG), echocardiogram (ECHO), vital signs, full hematology and biochemistry, Quality of Life questionnaire, radiologic assessments of baseline disease status and concomitant medications.

For patients with a history of liver surgery or major vasculature surgery, an angiogram evaluation of their vasculature will be performed for compatibility for Percutaneous Hepatic Perfusion (PHP) prior to confirming eligibility.

Eligibility date: This is the date on which all screening assessments have been completed and the patient is determined to be eligible for the trial.

Treatment Phase: Eligible patients will be treated with Melphalan/HDS 3.0 mg/kg Ideal Body Weight (IBW) and must begin treatment within 14 days being eligible. Melphalan/HDS treatment, patients will receive up to 6 treatments. Each treatment cycle consists of 6 weeks with an acceptable delay for another 2 weeks before the next planned treatment to allow for recovery of melphalan-related toxicity, if needed. Tumor response will be assessed every 12 weeks (+ 2 weeks) until disease progression. If the patient receives only 1 treatment, the disease assessment scans will be conducted 12 weeks after the date of the first treatment. The assessment scans will be reviewed by an Independent Review Committee (IRC), also referred to as Independent Central Review. At any time when progressive disease (PD) is observed, the patient will be removed from further study treatment and followed until death. Melphalan/HDS treatment will also be discontinued in the event that recovery from treatment related toxicity requires more than 8 weeks from last treatment. An end-of-treatment visit will be conducted approximately 6 to 8 weeks following the final study treatment. Ongoing treatment related adverse events (AEs) at the end-of-treatment visit will be followed until the severity is within one of the following parameters (1) Symptoms are resolved or return to baseline; (2) CTCAE Grade < 1 or can be explained; (3) patient death. The maximum possible duration of the study treatment for any patient will be 12 months.

NOTE: Active Melphalan/HDS patients (currently in treatment) on PHP-OCM-301 will continue treatment on PHP-OCM-301A following the re-consenting process.

NOTE: Patients on PHP-OCM-301 that have completed treatment and are entering or are already in the follow-up phase will be followed-up for survival and disease progression (as applicable) on PHP-OCM-301A following the re-consenting process.

Follow-up Phase: Once the patient has completed the end-of-treatment (EOT) visit in accordance with the schedule of events they will enter the follow-up phase. If the disease has not progressed at the EOT (Section 6.2), the patient will need to continue with disease assessment visits every 12 weeks (+ 2 weeks) until disease progression is documented. If the disease has progressed before or at the EOT their follow-up is to be by phone every 3 months for survival status until death.

Patients will be monitored, following the completion of study treatment, for the development of myelodysplasia and secondary leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. Patients must weigh ≥ 35 kg (due to possible size limitations with respect to percutaneous catheterization of the femoral artery and vein using the Delcath Hepatic Delivery System).
3. 50% or less histologically or cytologically-proven ocular melanoma metastases in the parenchyma of the liver.
4. Disease in the liver must be measurable by computed tomography (CT) and/or magnetic resonance imaging (MRI).
5. Evidence of limited extrahepatic disease on preoperative radiological studies is acceptable if the life threatening component of disease is in the liver. Limited extrahepatic disease is defined in this protocol as follows: metastasis in bone, subcutaneous, lung or lymph nodes that is amenable to resection or radiation and has a defined treatment plan. Patients with extra-hepatic tumor burden which does not have a defined treatment plan (i.e. monitor or is unable to be resected or radiated) must not be included in the trial.
6. Scans used to determine eligibility (CT scan of the chest/abdomen/pelvis and MRI of the liver) must be performed within 28 days prior to randomization. An MRI of the liver is required at screening to validate that CT accurately reflects the extent of disease in the liver. For patients with MRI intolerance, a 3-phase liver CT is to be done in place of liver MRI.
7. Patients must not have chemotherapy, radiotherapy, chemoembolization, radioembolization, or immunoembolization for their malignancy within 30 days prior to treatment and must have recovered from all side effects of therapeutic and diagnostic interventions except those listed in Appendix B of the study protocol.
8. Patients receiving anti programmed cell death protein 1 (PD-1) immunotherapy such as pembrolizumab or nivolumab, or human cytotoxic T-lymphocyte antigen 4 blocking antibody such as ipilimumab should wait 8 weeks before Melphalan/HDS treatment.
9. Patients must have an ECOG PS of 0-1 at screening and on the day prior to treatment.
10. Patients must have adequate hepatic function as evidenced by total serum bilirubin ≤ 1.5 x the upper limit of normal (ULN) and a prothrombin time (PT) within 2 seconds of the upper normal limit. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) must be ≤ 2.5 x ULN.
11. Patients must have a platelet count > 100,000/µL, hemoglobin ≥ 10.0 gm/dL, white blood cell count (WBC) > 2,000/uL, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, and a serum creatinine ≤ 1.5 mg/dL unless the measured creatinine clearance is > 40 mL/min/1.73 m2.
12. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (β-human chorionic gonadotropin) within 7 days prior to randomization.
13. Provided signed informed consent.

Exclusion Criteria:

1. Patients with Child-Pugh Class B or C cirrhosis or with evidence of portal hypertension by history, endoscopy, or radiologic studies.
2. Those with New York Heart Association functional classification II, III or IV active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
3. History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
4. Women of childbearing potential (WOCBP) i.e. fertile meaning not permanently sterilized and having had a menstrual period within the past 12 months) unable to undergo hormonal suppression to avoid menstruation during treatment.
5. WOCBP and fertile males (not permanently sterile by bilateral orchidectomy) unwilling or unable to use highly effective contraception method for consent to at least 6 months after the last administration of study treatment (e.g. combined hormonal contraception; progestogen-only hormonal contraception; Intrauterine device, intrauterine hormone-releasing system; bilateral tubal occlusion, vasectomized partner or sexual abstinence).
6. Females that are pregnant or breastfeeding patients
7. Patients taking immunosuppressive drugs; however, oral corticosteroids ≤ 10 mg/day are allowed.
8. Patients who are unable to be temporarily removed from chronic anti-coagulation therapy.
9. Patients with active bacterial infections with systemic manifestations (malaise, fever, leucocytosis) are not eligible until completion of appropriate therapy.
10. Patients with severe allergic reaction to iodine contrast, which cannot be controlled by premedication with antihistamines and steroids (because a hepatic angiogram is needed for the Delcath system procedure).
11. Patients with a history of or known hypersensitivity to melphalan or the components of the Melphalan/HDS system.
12. Patients with latex allergy.
13. Patients with a history of hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
14. Patients with a history of bleeding disorders or evidence of intracranial abnormalities which would put them at risk for bleeding with anti-coagulation (e.g., strokes, active metastases).
15. Patients with a history of gastrinoma, hepatic vasculature incompatible with perfusion, hepatofugal flow in the portal vein or known unresolved venous shunting.
16. Known varices at risk of bleeding, including medium or large esophageal or gastric varices, or active peptic ulcer.
17. Patients with prior Whipple's procedure.
18. Patients with brain metastases or presence of other intracranial lesions at risk for bleeding by history or baseline radiologic imaging.
19. Patients with active liver infection, including Hepatitis B and Hepatitis C infection. Patients with anti-hepatitis B core antibody (HBc) positive, or hepatitis B surface antigen (HBsAg) but DNA negative are exception(s).
20. Uncontrolled endocrine disorders including diabetes mellitus, hypothyroidism, or hyperthyroidism.
21. Received any investigational agent for any indication within 30 days prior to first treatment.
22. Not recovered from side effects of prior therapy to ≤ Grade 1 (according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v. 4.03). Certain side effects that are unlikely to develop into serious or life-threatening events (e.g. alopecia) are allowed at > Grade 1.
23. Cancers other than ocular melanoma for which the patient is currently under treatment or still deemed not to be cancer free.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as determined by Independent Central Review Committee | Patients will be assessed for ORR from baseline through completion of treatment. [assessed up to 36 months]
  ORR (complete or partial response)

SECONDARY OUTCOMES:
Duration of Response (DOR) as determined by Independent Central Review Committee | From time of 1st treatment until there is evidence of disease progression [assessed up to 36 months]
  Duration of Response (DOR) is defined as the time from first documented confirmed response of CR or PR based on RECIST v1.1 determined by the IRC to the first documented progression or death due to any cause.
Disease Control Rate (DCR) determined by Independent Central Review Committee | ORR will be assessed every 10-14 weeks from the start of 1st treatment and continues until the earlier of either when there is evidence of disease progression or 1 year from 1st treatment.
  DCR is defined as the proportion of patients with a best overall response of CR of any duration, PR of any duration, or stable disease (SD) for a minimum of 12 weeks from the eligibility date for PHP-OCM-301A patients (and randomization date for PHP-OCM-301 patients)
Overall Survival | From the start of the study to the date the patient was last known alive. [assessed up to 36 months]
  Overall Survival will be measured from the eligibility date for PHP-OCM-301A patients (and randomization date for PHP-OCM-301 patients) to the date of death (included all-cause mortality).
Progression-Free Survival | From start of study until disease progression. [assessed up to 36 months]
  PFS is defined as the time from the eligibility date for PHP-OCM-301A patients (and randomization date for PHP-OCM-301 patients) to the first occurrence of disease progression (either hepatic or extra-hepatic), as determined by the investigator and Independent Central Review Committee assessments using RECIST (version 1.1), or death from any cause.

OTHER OUTCOMES:
Time to Objective Response (TOR) | From study start through study completion. [Assessed up to 36 months]
  TOR will be summaries for each treatment group with descriptive statistics (n, median, quartiles, number censored, 95% confidence intervals, and hazard ratios) using Kaplan-Meier time-to-event analysis techniques.
The summary of ORR, DOR, DCR, PFS and TOR as determined from the Investigator-assessed objective response will follow the same approach as those determined by the IRC | Assessed from the start of 1st treatment and continues until there is evidence of disease progression or 1 year from 1st treatment.
  The ratio of patients with either a complete or partial response over the total of all patients in the study
Hepatic Progression Free Survival (hPFS) | Assessed from the start of study through evidence of hepatic disease progression [Assessed up to 36 months]
  Hepatic PFS (hPFS) is defined as the time from the eligibility date for the PHP-OCM-301A patients (and randomization date for PHP-OCM-301 patients) to the first occurrence of hepatic disease progression, as determined by the Independent Central Review Committee (IRC) on imaging studies using RECIST 1.1 or death from any cause.
Hepatic Objective Response Rate (hORR) as determined by Imaging Core Lab | Assessed from the start of 1st treatment and continues until there is evidence of disease progression in the liver or 1 year from 1st treatment. [Assessed up to 36 months]
  Hepatic Objective Response Rate (hORR), is defined as the proportion of patients with tumor size reduction when evaluating hepatic lesions after study treatment as determined by the IRC using RECIST version 1.1.
Quality of Life as Measured by Functional Hepatobiliary Symptom Index (FHSI-8) | Quality of life will be assessed at screening and last week of each treatment and at end of treatment, which is the earlier of either disease progression or 6-8 weeks after the last treatment. [Assessed over 12 months]
  Using a questionnaire, patients will self-assess how they feel after the treatment. A total of eight questions are to be answered, patients are asked to complete each question based on the previous 7 days. Rating of answers are 0 (not at all) up to 4 (very much). Questions are (1). if the patient has lack of energy, (2) does the patient have nausea, (3) does the patient have pain, (4) does the patient feel they are losing weight, (5) does the patient have back pain, (6) is the patient tired, (7) is the patient bother by jaundice or yellow coloring of skin, (8)does the patient have pain/discomfort in the stomach area, The FHSI-8 quality of life instrument will be scored per standard methodology developed for the questionnaire. Results will be presented by treatment groups; changes from baseline will also be calculated.
Exploratory Analysis for Demographics | From time of enrollment [assessed up to 24 months]
  Subgroup analysis of Demographic information, including age, gender, race, and ethnicity.
Exploratory analysis for the amount of liver involvement | From time of enrollment. [Assessed up to 24 months]
  Exploratory subgroup analyses will be performed by forming subsets of patients from the ITT population in order to evaluate the robustness of the results based on the primary efficacy analysis. These univariate analyses may include, but are not limited to, comparisons between treatment groups based on several baseline characteristics such as:
  • Extent of liver involvement (1-25% / 26-50%).
Exploratory Analysis of performance status | From study start to end of treatment. [Assessed up 36 months]
  Exploratory subgroup analyses will be performed by forming subsets of patients from the ITT population in order to evaluate the robustness of the results based on the primary efficacy analysis. These univariate analyses may include, but are not limited to, comparisons between treatment groups based on several baseline characteristics such as:
  • ECOG performance status (0,1 vs other)
Safety Outcome evaluation for Adverse Events | From the time of Informed consent through study completion. [assessed up to 36 months]
  All safety analyses will be based on the safety population. Summary statistics for continuous efficacy variables will include the mean, standard deviation, median and range (minimum/maximum).
Safety Outcome Evaluation of date for the development of Myelodysplasia and secondary leukemia | From the time of study completion until death. [Assessed up to 24 months]
  performed by forming subsets of patients from the ITT population in order to evaluate the robustness of the results based on the primary efficacy analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Zager, MD, Principal Investigator — Moffitt Cancer Center
Locations (24):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University James Cancer Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
- Universitätsklinikum Graz, Graz, Austria
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Centre Léon Bérard, Lyon, Rhône, France
- Germany (5):
  - Charité Unversitätsmedizin Berlin Comprehensive Cancer Center, Berlin
  - Universitätsklinikum Giessen und Marburg, Marburg
  - Universitätshautklinik Münster, Münster
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Würzburg, Würzburg
- Istituto Europeo di Oncologia, Milan, Italy
- Spain (2):
  - Clínic Barcelona, Barcelona
  - Hospital Ramón y Cajal, Madrid
- UniversitätsSpital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - University Hospital Southampton NHS Trust, Southampton, Hampshire
  - Aintree University Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zager JS, Orloff M, Ferrucci PF, Choi J, Eschelman DJ, Glazer ES, Ejaz A, Howard JH, Richtig E, Ochsenreither S, Reddy SA, Lowe MC, Beasley GM, Gesierich A, Bender A, Gschnell M, Dummer R, Rivoire M, Arance A, Fenwick SW, Sacco JJ, Haferkamp S, Weishaupt C, John J, Wheater M, Ottensmeier CH. Efficacy and Safety of the Melphalan/Hepatic Delivery System in Patients with Unresectable Metastatic Uveal Melanoma: Results from an Open-Label, Single-Arm, Multicenter Phase 3 Study. Ann Surg Oncol. 2024 Aug;31(8):5340-5351. doi: 10.1245/s10434-024-15293-x. Epub 2024 May 4. PMID 38704501